CLINICAL TRIAL: NCT03352362
Title: Comparison of the Effect of Propacetamol, Ibuprofen or Their Combination on Postoperative Pain and Quality of Recovery After Laparoscopic Hernia Repair in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4-2017-0869
Record Dates: First submitted 2017-11-20; First posted 2017-11-24 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal | interventions — Ibuprofen; propacetamol

STUDY DESIGN:
Intervention Model Description: Participants are divided 3 groups(caldolor, denogan, combination group) randomly. Each groups are received a medication by protocol during surgery
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- caldolor (Experimental): intravenous caldolor injection during intraoperative period
  Interventions: Drug: ibuprofen (caldolor 10 mg / kg)
- denogan (Active Comparator): intravenous denogan injection during intraoperative period
  Interventions: Drug: propacetamol (denogan 30 mg / kg)
- combination (Experimental): intravenous denogan and caldolor injection during intraoperative period
  Interventions: Drug: ibuprofen + propacetamol

INTERVENTIONS:
Drug: ibuprofen (caldolor 10 mg / kg) — Dilution caldolor 10 mg / kg in Hartmann solution to 50 mL - 100 mL and intravenous injection for 30 minutes immediately after induction of anesthesia
  Arms: caldolor
Drug: propacetamol (denogan 30 mg / kg) — Dilution denogan 30 mg / kg in the dissolved solution to a total of 10 ml and intravenous injection for 10 minutes after the main surgical procedure end
  Arms: denogan
Drug: ibuprofen + propacetamol — Dilution caldolor 10 mg / kg in Hartmann solution to 50 mL - 100 mL and intravenous injection for 30 minutes immediately after induction of anesthesia Dilution denogan 30 mg / kg in the dissolved solution to a total of 10 ml and intravenous injection for 10 minutes after the main surgical procedure end
  Arms: combination

SUMMARY:
There are difficulties in the progress of the study and cancel the plan. The purpose of this study is to evaluate the postoperative pain control using non - opioidal analgesics in children. The investigators will investigate the effect of single use and combination of caldorol(ibuprofen) compare to denogan(propacetamol) in children.

Participants who receive the laparoscopic inguinal hernia repair between 6 months and 6 years old are divided 3 groups(caldolor, denogan, combination). Each groups are received a medication by protocol during surgery. After operation patient's pain score and use of additional analgesics are recorded in postanesthesia care unit and general ward.

ELIGIBILITY:
Inclusion Criteria:

* scheduled to undergo laparoscopic inguinal hernia surgery
* American Society of Anesthesiologists physical status classification 1 or 2
* Children aged 6 months to 6 years

Exclusion Criteria:

* history of Gastrointestinal bleeding
* history or laboratory finding of suspected renal or hepatic dysfunction
* bronchial asthma
* bleeding disorder
* hypersensitivity to NSAID or propacetamol
* disagreement of investigation
* The researcher determines that participation is inappropriate due to other reasons.

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 159 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2019-03-08 (Actual); Study Completion 2019-03-09 (Actual)

PRIMARY OUTCOMES:
additional administration of analgesics | during stay time in PACU (postanesthesia care unit) average of over 30 minutes up to 1 hour
  whether additional analgesics are administered during the postanesthesia care unit due to pain

SECONDARY OUTCOMES:
pain score (FLACC) | Participant's pain score is evaluated by FLACC at the time of arriving the postanesthesia care unit(PACU)
  Face-legs-activity-cry-consolability scale(FLACC) - FLACC scale is a measurement used to assess pain for children between the ages of 2 months and 7 years or individuals that are unable to communicate their pain. The scale is scored in a range of 0-10 with 0 representing no pain. The scale has five criteria, which are each assigned a score of 0, 1 or 2.
pain score (FLACC) | Participant's pain score is evaluated by FLACC at 10 minutes after arriving the postanesthesia care unit(PACU)
  Face-legs-activity-cry-consolability scale(FLACC) - FLACC scale is a measurement used to assess pain for children between the ages of 2 months and 7 years or individuals that are unable to communicate their pain. The scale is scored in a range of 0-10 with 0 representing no pain. The scale has five criteria, which are each assigned a score of 0, 1 or 2.
pain score (FLACC) | Participant's pain score is evaluated by FLACC at 20 minutes after arriving the postanesthesia care unit(PACU)
  Face-legs-activity-cry-consolability scale(FLACC) - FLACC scale is a measurement used to assess pain for children between the ages of 2 months and 7 years or individuals that are unable to communicate their pain. The scale is scored in a range of 0-10 with 0 representing no pain. The scale has five criteria, which are each assigned a score of 0, 1 or 2.
pain score (FLACC) | Participant's pain score is evaluated by FLACC at the time of leaving the postanesthesia care unit(PACU) (up to 1 hour)
  Face-legs-activity-cry-consolability scale(FLACC) - FLACC scale is a measurement used to assess pain for children between the ages of 2 months and 7 years or individuals that are unable to communicate their pain. The scale is scored in a range of 0-10 with 0 representing no pain. The scale has five criteria, which are each assigned a score of 0, 1 or 2.
pain score (CHEOPS) | Participant's pain score is evaluated by FLACC at the time of arriving the postanesthesia care unit(PACU)
  Children's Hospital of Eastern Ontario Pain Scale(CHEOPS) - The CHEOPS is an observational scale for measuring postoperative pain in children aged 1-7 years. It can be used to monitor the effectiveness of interventions for reducing the pain and discomfort. It includes six categories of pain behavior, each with 3-4 levels and scores range from 4 points (no pain) to 13 points (the worst pain).
pain score (CHEOPS) | Participant's pain score is evaluated by FLACC at 10 minutes after arriving the postanesthesia care unit(PACU)
  Children's Hospital of Eastern Ontario Pain Scale(CHEOPS) - The CHEOPS is an observational scale for measuring postoperative pain in children aged 1-7 years. It can be used to monitor the effectiveness of interventions for reducing the pain and discomfort. It includes six categories of pain behavior, each with 3-4 levels and scores range from 4 points (no pain) to 13 points (the worst pain).
pain score (CHEOPS) | Participant's pain score is evaluated by FLACC at 20 minutes after arriving the postanesthesia care unit(PACU)
  Children's Hospital of Eastern Ontario Pain Scale(CHEOPS) - The CHEOPS is an observational scale for measuring postoperative pain in children aged 1-7 years. It can be used to monitor the effectiveness of interventions for reducing the pain and discomfort. It includes six categories of pain behavior, each with 3-4 levels and scores range from 4 points (no pain) to 13 points (the worst pain).
pain score (CHEOPS) | Participant's pain score is evaluated by FLACC at the time of leaving the postanesthesia care unit(PACU) (up to 1 hour)
  Children's Hospital of Eastern Ontario Pain Scale(CHEOPS) - The CHEOPS is an observational scale for measuring postoperative pain in children aged 1-7 years. It can be used to monitor the effectiveness of interventions for reducing the pain and discomfort. It includes six categories of pain behavior, each with 3-4 levels and scores range from 4 points (no pain) to 13 points (the worst pain).
pain score (PPPM scale) | The PPPM scale is measured at 4 hours after surgery
  Parents' Postoperative Pain Measure(PPPM scale): The number of items parents have circled "Yes" are summed for a total score out of 15. A score of at least 6 out of 15 signifies clinically significant pain.
pain score (PPPM scale) | The PPPM scale is measured at 12 hours after surgery
  Parents' Postoperative Pain Measure(PPPM scale): The number of items parents have circled "Yes" are summed for a total score out of 15. A score of at least 6 out of 15 signifies clinically significant pain.
pain score (PPPM scale) | The PPPM scale is measured at 24 hours after surgery
  Parents' Postoperative Pain Measure(PPPM scale): The number of items parents have circled "Yes" are summed for a total score out of 15. A score of at least 6 out of 15 signifies clinically significant pain.
incidence of complications | during stay time in PACU (postanesthesia care unit) average of over 30 minutes up to 1 hour
  incidence of complications in PACU (postanesthesia care unit)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain MedicineYonsei University College of Medicine Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee HM, Park JH, Park SJ, Choi H, Lee JR. Comparison of Monotherapy Versus Combination of Intravenous Ibuprofen and Propacetamol (Acetaminophen) for Reduction of Postoperative Opioid Administration in Children Undergoing Laparoscopic Hernia Repair: A Double-Blind Randomized Controlled Trial. Anesth Analg. 2021 Jul 1;133(1):168-175. doi: 10.1213/ANE.0000000000005284. PMID 33181557